CLINICAL TRIAL: NCT06866080
Title: An Open-label Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LCAR-AIO for the Treatment of Relapsed/Refractory Autoimmune Diseases (r/r AID)
Brief Title: A Study of LCAR-AIO in Subjects With Relapsed/Refractory Autoimmune Diseases
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Discontinue further development of LCAR-AIO program
Sponsor: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2305-0002
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Relapsed/Refractory Autoimmune Diseases
Keywords: Relapsed/Refractory Systemic lupus erythematosus (r/r SLE); Relapsed/Refractory Systemic Sclerosis (SSc); ), Relapsed/Refractory Anti-neutrophil cytoplastic antibodies (ANCA)-associated vasculitis (AAV); Idiopathic Relapsed/Refractory Inflammatory Myopathies (IIM)
MeSH Terms: conditions — Autoimmune Diseases; Recurrence; Lupus Erythematosus, Systemic; Scleroderma, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Myositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chimeric antigen receptor T cells (LCAR-AIO) (Experimental): Each subject will be given a single-dose LCAR-AIO cells infusion at each dose level
  Interventions: Biological: LCAR-AIO T cells

INTERVENTIONS:
Biological: LCAR-AIO T cells — Before treatment with LCAR-AIO T cells, subjects will receive a conditioning regimen.

SUMMARY:
This is a prospective, single-arm, open-label, dose-exploration and expansion clinical study of LCAR-AIO in adult subjects with relapsed/refractory autoimmune diseases.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label exploratory clinical study to evaluate the safety, tolerability, pharmacokinetics and efficacy profiles of LCAR-AIO, a chimeric antigen receptor (CAR) -T cell therapy in subjects with relapsed/refractory autoimmune diseases. Patients who meet the eligibility criteria will receive LCAR-AIO infusion. The study will include the following sequential stages: screening, apheresis, pre-treatment (cell product preparation: lymphodepleting chemotherapy), treatment (LCAR AIO infusion) and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in clinical research.
2. Age 18-65 years.
3. Adequate organ function at screening.
4. Clinical laboratory values meet criteria at screening.

SLE:

* Have been diagnosed of SLE at least 6 months before screening.
* At screening, antinuclear antibody, and/or anti-dsDNA antibody, and/or anti-Smith antibody should be positive.
* Fulfill relapsed/refractory SLE conditions.

AAV:

* Have been diagnosed of AAV before screening.
* Positive test for anti-PR3 or anti-MPO antibodies at screening.
* Fulfill relapsed/refractory AAV conditions.

SSc:

* Have been diagnosed of SSc before screening.
* At screening, mRSS is higher than 10.
* Fulfill relapsed/refractory SSc conditions.

IIM:

* Have been diagnosed of IIM before screening.
* Positive test for myositis-associated antibodies or myositis-specific antibodies at screening.
* Fulfill relapsed/refractory IIM conditions.

Exclusion Criteria:

1. Active infections such as hepatitis and tuberculosis.
2. Other autoimmune diseases.
3. Serious underlying diseases such as tumor, uncontrolled diabetes.
4. Female subjects who were pregnant, breastfeeding, or planning to become pregnant while participating in this study or within 1 year of receiving LCAR-AIO treatment.
5. Participated in other clinical trials within 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Change in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) scores from baseline up to 104 weeks | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  • The SLEDAI-2K scale is a cumulative and weighted index used to assess disease activity across 24 different disease descriptors in patients with SLE. A total score can fall between 0 and 105, with a higher score representing a more significant degree of disease activity.
Change in Birmingham vasculitis activity score (BVAS) from baseline up to 104 weeks | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  • The BVAS is a cumulative and weighted index used to assess disease activity across 9 organ systems in patients with AAV. A total score can fall between 0 and 64, with a higher score representing a more significant degree of disease activity.
Change in modified Rodnan skin score (mRSS) from baseline up to 104 weeks | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  • The mRSS is a scale used to assess skin thickness and scope of SSc patients by physically evaluating 17 positions. A total score can fall between 0 and 51, with a higher score representing a more significant degree of skin involvement.
Change in manual muscle testing (MMT-8) score from baseline up to 104 weeks | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  • This validated tool assesses muscle strength through muscle testing an abbreviated group of 8 proximal, distal, and axial muscles in IIM patients. A total score can fall between 0 and 150, with a lower score representing a more significant degree of muscle involvement.
Change in Physician global assessment (PGA) scores from baseline up to 104 weeks | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  • The physician will evaluating the global activity of AID patients by placing a vertical line on a 100-mm visual analog scale on which the left-hand boundary represents "no activity", and the right-hand boundary represents "the most severe activity".
Changes from baseline in immunological markers and Immunogenicity (anti-drug antibody) from baseline up to 104 weeks | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  • Detection of Immunoglobulins, autoantibodies (anti-dsDNA antibody, anti-Smith antibody, etc.) and anti-drug antibody.

SECONDARY OUTCOMES:
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  • An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment.
Incidence of dose-limiting toxicity (DLT) | 30 days after LCAR-AIO infusion (Day 1)
  • DLTs are severe adverse events refers to any untoward medical occurred in a subject participated in a clinical investigation, which have a causal relationship with the treatment and will limit the dose escalation.
Pharmacokinetics in peripheral blood | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  • CAR positive T cells levels in peripheral blood after LCAR-AIO infusion.
Recommended Dose regimen finding | Maximum 104 Weeks after LCAR-AIO infusion (Day 1)
  Recommended Dose regimen established through dose exploratory.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First Affiliated Hospital of USTC (anhui provincial hospital), Hefei
  - Jiangsu Province Hospital, Nanjing
  - The 1st Affiliated Hospital of WHU, Wenzhou
  - The Affiliated Hospital of XUZHOU Medical University, Xuzhou

IPD SHARING:
Plan to Share IPD: No